CLINICAL TRIAL: NCT04239937
Title: Insulin Resistance in Stress-metabolic Medical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Slagelse Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-800
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Septic Shock; Sepsis; Insulin Resistance
MeSH Terms: conditions — Shock, Septic; Sepsis; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study on the insulin resistance in sepsis and septic shock patients.

DETAILED DESCRIPTION:
This observational study is inspired by the short-term insulin resistance and hyperglycemia that have been demonstrated in post-operative patients in response to tissue injury by Van den Berghe et al 2001. This short-term insulin resistance and hyperglycemia have also been observed in acutely ill patients (Van den Berghe et al 2006). The underlying mechanism for why acute ill patients have short-term insulin resistance is still unclear, but it is believed that the basic mechanism is increased glucose regeneration and gluconeogenesis, which is the consequence of stress metabolism. Hyperglycemia can occur as a result of insulin resistance and is associated with an increased risk of multiple complications, which is why it is important to detect and treat (Van den Berghe et al 2001). This also means that the more insulin-resistant the patient has been prior to the acute condition, the greater the risk of elevated blood glucose concentrations. PRS Review Comments identify apparent errors, deficiencies, or inconsistencies in the submitted information. Any comments provided should not be considered comprehensive. Advisory comments noted in a previous version of a study record may apply to subsequent versions, even if not repeated. It is the responsibility of the data provider to ensure that the record is consistent with the ClinicalTrials.gov Review Criteria.

The aim of the study is to clarify the degree of insulin resistance in medical patients who are not diagnosed with diabetes. Further it will be clarified how long these patients remain insulin resistant after discharge.

The acute medical patients diagnosed with sepsis or septic shock will be observed during hospitalization and after discharge. Sepsis is defined as life-threatening organ dysfunction caused by dysregulated host response to infection. Because the entire body is affected by an infection, it is expected that this group of patients have a high level of stress metabolism, insulin resistance and increased gluconeogenesis. The hypothesis is that acute medical patients diagnosed with sepsis or septic shock have a level of insulin resistance (days to weeks) and thus an increased risk of hyperglycemia. Insulin resistance is expected to decrease as the patient's condition improves.

The hypothesis is:

Patients with elevated infection levels (CRP and leukocyte count) who are simultaneously diagnosed with sepsis, has peripheral insulin resistance due to stress metabolism.

The pancreas will try to compensate for the peripheral insulin resistance by increasing its secretion of insulin to the bloodstream. C-peptide is excreted in equimolar amounts to insulin, thereby C-peptide becomes an expression of peripheral insulin resistance.

It is assumed that the insulin resistance gradually decreases after discharge and further as the patient's condition improves (CRP and leukocyte counts).

The study design is a prospective follow-up study. The difference in C-peptide will be observed over a time period of 28 days as an expression of the participant's insulin secretion. Futher, the participants' blood glucose will also be observed continuously to find the correlation between the degree of insulin resistance and glucose concentration. In addition, measure the correlation between the degree of infection and the increase in C-peptide concentration.

The primary endpoint is the change in C-peptide (the difference between the maximum concentration and the concentration after 28 days).

Secondary endpoints:

* The area under the curve for blood glucose level measured over 28 days.
* Correlation of infection level (CRP/leukocyte count) and increase in C-peptide concentration (dose-response).
* Correlation between infection rate and insulin resistance.

Patients admitted to the hospital with sepsis or septic shock can be recruited. Patients will be followed for 28 days from admission. The patients will be applied to a continuous flash glucose monitor (FGM) on the first day. Follow-up will be performed by blood sampling of C-peptide, leukocyte count, and CRP. HbA1c will also be measured for the exclusion of diabetes. Blood sampling will be taken both during hospitalization and after discharge. C-peptide will be measured every second day during hospitalization and leukocyte count and CRP will be measured every day during hospitalization. Reading of FGM will be performed on the 14. and on the 28. day where blood sampling of C-peptide, leukocyte count, and CRP also will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis or septic shock who are admitted to the emergency ward and subsequently transferred to an intensive, intermediate or medical ward at Slagelse Hospital. Patients are diagnosed with sepsis or septic shock based on screening using Sequential (sepsis-related) Organ Failure Assessment (SOFA) or Quick SOFA (qSOFA).
* Patients must be of legal age.

Exclusion Criteria:

* Patients with diabetes (T1DM or T2DM)
* Patients with terminal cancer
* Patients who are already participating in a trial
* Patients who do not understand and speak danish
* Patients who are demented
* Postoperative patients <1 month after surgery
* Patients who are going through dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sepsis or septic shock patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-08-27 (Estimated); Study Completion 2020-08-27 (Estimated)

PRIMARY OUTCOMES:
C-peptide | 28 days
  Changes in C-peptide over time

SECONDARY OUTCOMES:
Blood glucose level | 28 days
  The area under the curve for blood glucose level measured over 28 days
Infection level and C-peptide concentration | 28 days
  Correlation of infection level (CRP/leukocyte count) and increase in C-peptide concentration (dose-response).
Correlation between infection rate and insulin resistance. | 28 days
  Correlation between infection rate and insulin resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Slagelse Hospital, Slagelse, Denmark